CLINICAL TRIAL: NCT04352621
Title: Ketamine Enhancement of rTMS for Refractory Depression
Brief Title: Study to Assess the Effects of Intranasal Ketamine Along With rTMS for Patients With Treatment-resistant Major Depressive Disorder (TRD)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Erik Nelson, MD, Associate Professor, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nelson Ketamine IIT
Record Dates: First submitted 2020-02-16; First posted 2020-04-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Major Depressive Disorder
Keywords: treatment-resistant major depressive
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Ketamine; Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: To assess the effects of 0.5 mg/kg intranasal ketamine on response to rTMS treatment as measured by the Inventory for Depressive Symptomatology, Self-Rated Version (IDS-SR) in patients with treatment resistant depression (< 25% response to between 1 and 4 adequate antidepressant trials in the current episode).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ketamine plus rTMS (Experimental): Patients will be given a dose of ketamine followed by 6 weeks of rTMS treatment.
  Interventions: Drug: intranasal ketamine; Device: rTMS treatment

INTERVENTIONS:
Drug: intranasal ketamine — Ketamine 0.5 mg/kg will be administered intranasally using an atomization device with a maximum dose of 40 mg followed by 6 weeks of rTMS treatment. .
  Other Names: Ketamine
Device: rTMS treatment — patients will begin the open label trial of rTMS per the FDA-approved method on day 1 (the day after the Baseline Visit).
  Other Names: Repetitive transcranial magnetic stimulation (rTMS)

SUMMARY:
An open label study to assess the safety, tolerability, and effects of intranasal Ketamine in combination with rTMS for patients with treatment-resistant major depressive disorder (TRD). Patients will be given a dose of ketamine followed by 6 weeks of rTMS treatment.

DETAILED DESCRIPTION:
Investigate the effects of pretreatment using a single, sub-anesthetic dose of intranasal ketamine on the response to a standard course of rTMS in patients who meet the definition of TRD.

ELIGIBILITY:
Inclusion Criteria:

1. Males and non-pregnant females currently meeting the DSM-5 criteria for diagnosis of major depressive disorder (MDD), single episode or recurrent, with a current episode duration of 3 years or less (confirmed with the MINI);
2. episode has a Clinical Global Impressions Severity of Illness (CGI-S) score of at least 4 and a total score of at least 20 on the 17-item Hamilton Depression Rating Scale (HAMD17)
3. Age between 18-65
4. HAMD17 total score of at least 20 and a decrease in score of 25% or less from that observed at the screening assessment
5. Willing and able to provide informed consent
6. History of failure to respond (<25% improvement) to at least one, but not more than four antidepressant trial in the current episode. Alternatively, patients will be eligible if they have marked intolerance to antidepressants as demonstrated by four failed attempts to tolerate an adequate medication trial (lifetime).

Exclusion Criteria:

1. Unable to speak English well enough to participate in the rating scales which will only be provided in English.
2. Pregnancy or lactation
3. Post-partum state (within 2 months of delivery);
4. History of substance abuse or dependence within the past year (except nicotine and caffeine)
5. a lifetime history of psychosis, bipolar disorder, or obsessive- compulsive disorder;
6. diagnosis of posttraumatic stress disorder or an eating disorder in the past year
7. lack of response to a past adequate trial of electroconvulsive therapy (ECT) for MDD;
8. prior treatment with TMS or a vagus nerve stimulator implant;
9. use of hallucinogen in the last month
10. Current treatment with any medication NMDA receptor effects
11. Any history of prior ketamine use
12. Any clinically-significant medication or condition that would preclude the use of ketamine.
13. History of: a dissociative disorder, seasonal patteren of depression as defined by DSM-IV, any condition likely to be associated with increased intracranial pressure, space occyping lesion, seizure disorder except childhood febrile seizures, neurologic disorder or medication therapy known to alter seizure threshold, cerebrovascular accident, transient ischemic attack within the last 2 years, cerebral aneurysm, dementia, parkinson's disease, hunging's disease, multiple sclerosis, or a personality disorder (which in the judgement of the Investigator may hinder the patient in completing the procedures required by the study protocol)
14. Presence of ferromagnetic material in or in close proximity to the head.
15. Increased risk of seizure for any other reason, including prior diagnosis of increased intracranial pressure, pseudotumor cerebri, or history of significant head trauma with loss of consciousness for greater than or equal to 5 minutes
16. A true positive response to any question on the Transcranial Magnetic Stimulation Adult Safety Screen questionnaire
17. Inability to locate and quantify a motor threshold as defined in the protocol
18. ECT treatment within 3 months prior to the screening visit
19. Use of any investigational drug within 4 weeks of the baseline visit
20. Use of fluoxetine within 6 weeks of the baseline visit
21. Use of an MAOI within 2 weeks of the baseline visit
22. Use of any antidepressant within 1 week of the baseline visit
23. Significant acute suicide risk, defined as follows: Suicide attempt within the previous 6 months that required medical treatment; or Greater than or equal to 2 suicide attempts in the past 12 months; or
24. Has a clear-cut plan for suicide and states that he/she cannot guarantee that he/she will call his/her regular psychiatrist or the Investigator if the impulse to implement the plan becomes substantial during the study; or In the investigator's opinion, is likely to attempt suicide within the next 6 months.
25. Cardiac pacemakers, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease;
26. If participating in psychotherapy, must have been in stable treatment for at least 3 months prior to entry into the study, with no anticipation of change in the frequency of therapeutic sessions, or the therapeutic focus over the duration of the rTMS trial
27. Positive urine drug screen. (A positive urine drug screen at screening may be repeated once prior to randomization)
28. Clinically significant laboratory abnormality on CBC, TSH, ECG or hepatic profile in the opinion of the Investigator
29. Any known hypersensitivity or serious adverse effect with ketamine
30. Any clinically-significant medication or condition that would preclude the use of ketamine including respiratory illness requiring the regular use of oxygen.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Inventory for Depressive Symptomatology - Self-Rated | Screening to through study completion, an average of 42 days
  To assess the effects of 0.5 mg/kg intranasal ketamine on response to rTMS treatment as measured by the Inventory for Depressive Symptomatology, Self-Rated Version (IDS-SR) in patients with strictly defined treatment resistant depression.

IPD SHARING:
Plan to Share IPD: No